CLINICAL TRIAL: NCT05029492
Title: Effect of Visceral Manipulation on Polycystic Ovarian Syndrome
Brief Title: Effect of Visceral Manipulation on PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahitab Mohammed Yosri Ibrahim (Other)
Responsible Party: Sponsor-Investigator, Mahitab Mohammed Yosri Ibrahim, Lecturer of physical therapy for women's health, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/001044
Record Dates: First submitted 2021-08-15; First posted 2021-08-31 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Menstruation Disturbances; Caloric Restriction; Manipulation Therapy
MeSH Terms: conditions — Polycystic Ovary Syndrome; Menstruation Disturbances | interventions — Caloric Restriction; Control Groups; Population Groups; Diet

STUDY DESIGN:
Intervention Model Description: Polycystic ovarian women were assigned to either group (A), receiving a low-calorie diet for three months, or group (B), receiving the same diet as group (A) together with visceral manipulation of the pelvic organs and their related structures for the same study period (three months).
Who Masked: Outcomes Assessor
Masking Description: an independent researcher assigned the participants to one of the two study groups, by opening sealed envelopes containing serially ordered numbers. An independent assessor analyzed the patients' blood samples for hormonal profile and another assessor blinded to patients' allocation interviewed the patients for the questionnaire and assessed the weight.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet group (Active Comparator): Giving a low caloric diet
  Interventions: Other: Low-calorie diet
- Visceral manipulation with diet group (Experimental): Giving visceral manipulation added to a low-calorie diet
  Interventions: Other: Visceral manipulation with diet

INTERVENTIONS:
Other: Low-calorie diet — Low-calorie diet of 1200 kcal for 3 months, modified every two weeks.
  Other Names: Control group; Group (A)
  Arms: Diet group
Other: Visceral manipulation with diet — Visceral manipulation to the pelvic organs and their related structures (8 sessions, once per week in the first month then once every other week for two months) added to the same low-calorie diet as the group (A).
  Other Names: Study group; Group (B)
  Arms: Visceral manipulation with diet group

SUMMARY:
The study was conducted to determine the effect of visceral manipulation on menstrual irregularities and hormonal profile in women with polycystic ovarian syndrome. Thirty women were randomly and equally assigned into the group (A) (Control group), who received a low caloric diet (1200 Kcal/day) only for 3 months, and the group (B) (Study group), who received visceral manipulation to the pelvic organs and the related structures in addition to the same low-calorie diet as the group (A). Evaluations pre and post-study were done for body weight, BMI, female reproductive hormones, and menstruation-related problems.

DETAILED DESCRIPTION:
The current study was conducted to determine the effect of visceral manipulation on menstrual irregularities and hormonal profile in women with polycystic ovarian syndrome (PCOS). Thirty women having PCOS were chosen from the outpatient clinic of the faculty of physical therapy, Cairo University. Patients were randomly assigned into two groups equal in number. Group (A) (Control group), 15 PCOS women received a low caloric diet (1200 Kcal/day) for 3 months, while group (B) (Study group), 15 PCOS women received visceral manipulation to the pelvic organs and the related structures (8 sessions, once per week in the first month then once every other week for two months) in addition to the same low-calorie diet as the group (A). Evaluations pre and post-study for body weight, body mass index, female reproductive hormones [luteinizinghormone (LH), follicle-stimulating hormone (FSH) and LH/FSH ratio] and menstruation-related problems were done by weight- height scale, blood analysis, and menstruation-specific domain of polycystic ovary syndrome health-related quality of life questionnaire (PCOSQ), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Women having PCOS.
* 25 ≤ BMI ≤ 30 Kg/m2.
* Waist/hip ratio ≤ 0.80.
* Women experiencing irregular menstrual cycles.

Exclusion Criteria:

* Having cardiovascular diseases, diabetes mellitus, and/ or hypertension
* Having malignancy.
* Presence of reproductive disorders unrelated to PCOS.
* Presence of adrenal gland abnormalities.

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change of menstrual complaints' severity | At baseline and after three months of the intervention.
  The total score of menstruation- specific domain of polycystic ovarian syndrome questionnaire (PCOSQ) questions, calculated using the following equation: Number of patient/ group x number of questions/ domain. That total score was then used to determine the percentage of change from severity towards the optimal function.

SECONDARY OUTCOMES:
Change in the levels of reproductive hormones (FSH, LH, LH/FSH ratio) | At baseline in the second day of menstruation and after three months of the intervention.
  Human LH and FSH enzyme linked immunosorbent assay (ELISA) kits were used to assess the level of LH and FSH in the blood sample taken from each patient.
Change in weight | At baseline and after three months of the intervention.
  A weight- height scale is used to assess body weight in kilograms.
Change in Body mass index (BMI) | At baseline and after three months of the intervention.
  BMI is measured by the equation weight (Kg)/ height (m^2)

CONTACTS AND LOCATIONS:
Overall Officials: Mahitab Yosri, Lecturer of women's health, Principal Investigator — Cairo University